CLINICAL TRIAL: NCT02493166
Title: Cognitive Motor Interference During Dual Tasking With Movements of the Upper Limb in Persons With Multiple Sclerosis
Brief Title: Dual Task Cost in the Upper Limb in Persons With Multiple Sclerosis
Acronym: DTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: AZ Klina (Other); University Hospital, Antwerp (Other); private practice physician De Barsy (Unknown)
Responsible Party: Principal Investigator, Peter Feys, prof. dr., Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015-PFE-JRA01
Record Dates: First submitted 2015-07-02; First posted 2015-07-09 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with Multiple sclerosis Dual task cost (Active Comparator): Dual task cost (cognitive-motor interference), comparing single versus dual task performance (on both motor and cognitive task)
  Interventions: Other: dual task cost (cognitive-motor interference)
- Healthy volontiers Dual task cost (Active Comparator): Dual task cost (cognitive-motor interference), comparing single versus dual task performance (on both motor and cognitive task)
  Interventions: Other: dual task cost (cognitive-motor interference)

INTERVENTIONS:
Other: dual task cost (cognitive-motor interference) — comparing single versus dual task performance (on both motor and cognitive task)

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory, neurodegenerative disorder of the central nervous system, with more than 2.5 million people in the world. It is the most non-traumatic cause of disability in young and middle-aged adults.

Because the lesions are spread in the brains, there is a variety of symptoms. The most common symptom is the typical motor dysfunction. 66% of persons with MS, and even 81% of them after 15 years, have problems with movements in one or both upper extremities.

Also, 40 untill 70% of persons with Multiple Sclerosis have cognitive impairment. Although they are less visible, they can have a major determining influence on social or work-related domains. The most frequent cognitive dysfunctions are sustained attention, reduced speed of information processing, impaired memory and limited executive functions.

When a combination, of motor and cognitive task, is asked, the execution of these tasks could be difficult with the foregoing in mind. For example problems during chatting while cooking, typing a report at a meeting or watching television while ironing.

The dual-task paradigm assumes that the attention should be divided between two simultaneous tasks. A dual task cost (DTC) is a restriction in performance on each task, compared whit the separate task versus simultaneously.

Research on dual tasking with persons with MS has already studied extensively, but not specific on the upper limb. In 2015 Learmonth, Pilutti and Motl published an primary research on the DTC. They combined the movements of the upper limb with a cognitive task. The research showed a difference between Persons with MS and the control group. At methodological level, there is lacking on the randomization of tasks. That is an important bias because of the learning effect of the tasks. They used only one task for the upper limb; this isn't enough to generalize the concept of motor interference in Persons with MS.

The study has two research questions:

* Have Persons with MS a greater DTC compared with a healthy control group? The motor task is executed with the upper limb.
* Is there a difference on DTC in persons with MS depending on the motor task?

This research is an observational case-control study in which individuals with MS will be compared to a healthy control group. They will be two moments of assessments. On the first day the general performance of the persons will be measured, by using clinical evaluation tests and questionnaires. On the second day they will be tests on the dual tasks, specific a comparison between single versus simultaneously performed tasks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to McDonald's criteria
* 18+
* Have no other neurological or orthopedic disorder of the upper limb or spine. They should have the possibility to actively participate in the research.
* Nine hole peg test, in which the cut-off value is set at 0.5 PEG / sec

Exclusion Criteria:

* Patients are excluded with serious psychological problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
single motor task cost | day 1
  comparing single versus dual task performance on motor task
Dual motor task cost | day 2
  Comparing single versus dual task performance on congnitive task
single cognitive task cost | day 1
  Comparing single versus dual task performance on congnitive task
Dual cognitive task cost | day 2
  Comparing single versus dual task performance on congnitive task

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Joke Raats, Study Chair — AZ Klina
Locations (4):
- Belgium (4):
  - AZ Klina, Brasschaat
  - Private practice physician De Barsy, Brasschaat
  - Hasselt University, Diepenbeek
  - UZ Antwerp, Edegem